CLINICAL TRIAL: NCT01859806
Title: Isolated Roux Loop Pancreaticojejunostomy Versus Pancreaticogastrostomy After Pancreaticoduodenectomy
Acronym: PD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ayman El Nakeeb, Ass. Prof., Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pancreatic anastomosis
Record Dates: First submitted 2013-05-14; First posted 2013-05-22 (Estimated); Last update posted 2013-05-22 (Estimated); Status verified 2011-01

CONDITIONS: Pancreatic Fistula After Pancreaticoduodenectomy
Keywords: periampullary tumour; isolated Roux loop PJ; PG

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pancreaticogastrostomy group (Active Comparator): Standard PD with regional lymphadenectomy was performed. PG was done between pancreatic stump and posterior surface of the stomach with 2 layer interrupted anastomosis,and duct to mucosa.
  Interventions: Procedure: Pancreaticogastrostomy group
- Isolated Roux PJ group (Active Comparator): Isolated Roux PJ group, reconstruction was begun using the transected jejunum and ,which was anastomosed in end to side fashion. A separate Roux loop was performed for HJ, by dividing the jejunum about 40 cm beyond the pancreatic anastomosis and GJ was done in this loop (30 cm caudally from HJ). The PJ loop was anastomosed to the main loop (20 cm caudal to GJ).
  Interventions: Procedure: Isolated Roux PJ group

INTERVENTIONS:
Procedure: Pancreaticogastrostomy group — Standard PD with regional lymphadenectomy was performed. PG was done between pancreatic stump and posterior surface of the stomach with 2 layer interrupted anastomosis,and duct to mucosa.
  Other Names: Group 1
  Arms: Pancreaticogastrostomy group
Procedure: Isolated Roux PJ group — Isolated Roux PJ group, reconstruction was begun using the transected jejunum and ,which was anastomosed in end to side fashion. A separate Roux loop was performed for HJ, by dividing the jejunum about 40 cm beyond the pancreatic anastomosis and GJ was done in this loop (30 cm caudally from HJ). The PJ loop was anastomosed to the main loop (20 cm caudal to GJ).
  Other Names: Group 2
  Arms: Isolated Roux PJ group

SUMMARY:
Pancreaticoduodenectomy (PD)is the treatment of choice for patients with periampullary tumour (benign or malignant). In the recent years, the mortality rate of PD has decreased to 5% in many centers. However, pancreatic fistula (POPF) still occurs in 5 % to 40% of patients after PD. The hypothesis that isolated Roux loop PJ with isolated pancreatic drainage decrease the incidence of PF and severity with preservation of pancreatic function.

So the investigators compare isolated Roux Loop Pancreaticojejunostomy (PJ) Versus Pancreaticogastrostomy (PG) as regards incidence of POPF, severity of POPF and functional outcome.

DETAILED DESCRIPTION:
The hypothesis that isolated Roux loop PJ decrease the incidence of PF and severity with preservation of pancreatic function (exocrine and endocrine functions).

Preoperative evaluation included abdominal CT, liver function, tumor marker CEA, CA19-9, preoperative ERCP were optional in selected cases (patients with high bilirubin with high enzymes. Patients with distant metastasis or locally advanced were excluded.

Informed consent was obtained from all patients entered in the study Randomization: enrolled patients were randomized intraoperatively after PD resection to either isolated Roux PJ with isolated pancreatic drainage group or PG group by closed envelope which withdrawn by the nurse.

Operative technique. Standard PD with regional lymphadenectomy was performed. PG was done between pancreatic stump and posterior surface of the stomach with 2 layer interrupted anastomosis,and duct to mucosa.

Isolated Roux PJ group, reconstruction was begun using the transected jejunum and, which was anastomosed in end to side fashion. A separate Roux loop was performed for HJ, by dividing the jejunum about 40 cm beyond the pancreatic anastomosis and GJ was done in this loop (30 cm caudally from HJ). The PJ loop was anastomosed to the main loop (20 cm caudal to GJ).

One intrabdominal drains in morrison space. Intraoperative data and postoperative data were collected. Pancreatic function assessment.

The primary outcome was assessment the incidence of POPF after isolated Roux PJ and PG. The secondary outcomes were intraoperative blood loss, drain amount,day to resume oral intake hospital stay, operative duration, pancreatic function, postoperative complications delayed gastric emptying,

ELIGIBILITY:
Inclusion Criteria:

* All periampullary tumour either benign or resectable malignant tumour

Exclusion Criteria:

* locally advanced tumour infiltrating SMA
* Metastasis
* unfit

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2011-01; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Postoperative pancreatic fistula (POPF) | one year postoperative
  Postoperative pancreatic fistula was defined as drainage of > 50 ml/d of amylase rich fluid( 3 folds elevation above upper limit of normal in serum)

SECONDARY OUTCOMES:
Pancreatic function | one year postoperative
  Steatorrhea, blood glucose, fat in stool
Postoperative complications | one year postoperative
  Delayed gastric emptying, bile leakage, bleeding PG, bleeding GJ
Operative duration | 8 hours
  Operative duration
hospital stay | 5 weeks
  hospital stay,

CONTACTS AND LOCATIONS:
Overall Officials: Ayman El Nakeeb, MD, Principal Investigator — Mansoura University
Locations (1):
- Ayman El Nakeeb, Al Mansurah, Mansoura, Egypt

REFERENCES:
- [Background] Sutton CD, Garcea G, White SA, O'Leary E, Marshall LJ, Berry DP, Dennison AR. Isolated Roux-loop pancreaticojejunostomy: a series of 61 patients with zero postoperative pancreaticoenteric leaks. J Gastrointest Surg. 2004 Sep-Oct;8(6):701-5. doi: 10.1016/j.gassur.2004.05.001. PMID 15358331
- [Background] El Nakeeb A, Salah T, Sultan A, El Hemaly M, Askr W, Ezzat H, Hamdy E, Atef E, El Hanafy E, El-Geidie A, Abdel Wahab M, Abdallah T. Pancreatic anastomotic leakage after pancreaticoduodenectomy. Risk factors, clinical predictors, and management (single center experience). World J Surg. 2013 Jun;37(6):1405-18. doi: 10.1007/s00268-013-1998-5. PMID 23494109
- [Result] Ballas K, Symeonidis N, Rafailidis S, Pavlidis T, Marakis G, Mavroudis N, Sakantamis A. Use of isolated Roux loop for pancreaticojejunostomy reconstruction after pancreaticoduodenectomy. World J Gastroenterol. 2010 Jul 7;16(25):3178-82. doi: 10.3748/wjg.v16.i25.3178. PMID 20593503
- [Result] Kaman L, Sanyal S, Behera A, Singh R, Katariya RN. Isolated roux loop pancreaticojejunostomy vs single loop pancreaticojejunostomy after pancreaticoduodenectomy. Int J Surg. 2008 Aug;6(4):306-10. doi: 10.1016/j.ijsu.2008.04.007. Epub 2008 May 8. PMID 18556251
- [Result] Fragulidis GP, Arkadopoulos N, Vassiliou I, Marinis A, Theodosopoulos T, Stafyla V, Kyriazi M, Karapanos K, Dafnios N, Polydorou A, Voros D, Smyrniotis V. Pancreatic leakage after pancreaticoduodenectomy: the impact of the isolated jejunal loop length and anastomotic technique of the pancreatic stump. Pancreas. 2009 Oct;38(7):e177-82. doi: 10.1097/MPA.0b013e3181b57705. PMID 19730152
- [Result] Kingsnorth AN. Safety and function of isolated Roux loop pancreaticojejunostomy after Whipple's pancreaticoduodenectomy. Ann R Coll Surg Engl. 1994 May;76(3):175-9. PMID 7912489
- [Result] Khan AW, Agarwal AK, Davidson BR. Isolated Roux Loop duct-to-mucosa pancreaticojejunostomy avoids pancreatic leaks in pancreaticoduodenectomy. Dig Surg. 2002;19(3):199-204. doi: 10.1159/000064213. PMID 12119522
- [Result] Ke S, Ding XM, Gao J, Zhao AM, Deng GY, Ma RL, Xin ZH, Ning CM, Sun WB. A prospective, randomized trial of Roux-en-Y reconstruction with isolated pancreatic drainage versus conventional loop reconstruction after pancreaticoduodenectomy. Surgery. 2013 Jun;153(6):743-52. doi: 10.1016/j.surg.2013.02.008. Epub 2013 Apr 16. PMID 23601899
- See also: Mansoura university, Mansoura, Egypt — http://www.mans.edu.eg/